CLINICAL TRIAL: NCT04732910
Title: CFTR Biomarker Studie Bei Patient*Innen Mit Mukoviszidose Und CFTR-Modulatortherapie
Brief Title: Cystic Fibrosis Transmembrane Regulator (CFTR) Biomarker Study to Evaluate the Rescue of Mutant CFTR in Patients With Cystic Fibrosis Treated With CFTR-modulators
Acronym: Modulate-CF
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hannover Medical School (Other); Heidelberg University (Other); University of Giessen (Other)
Responsible Party: Principal Investigator, Simon Graeber, BIH Clinician Scientist, Charite University, Berlin, Germany
Other Study IDs: 20012746
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
Keywords: CFTR; ICM; NPD
MeSH Terms: conditions — Cystic Fibrosis | interventions — Therapeutics; lumacaftor, ivacaftor drug combination; tezacaftor, ivacaftor drug combination; elexacaftor, ivacaftor, tezacaftor drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Treatment with cystic fibrosis transmembrane regulator (CFTR) modualtors Ivacaftor, Lumacaftor-Ivacaftor, Tezacaftor-Ivacaftor, Elexacaftor-Tezacaftor-Ivacaftor — observational

SUMMARY:
This observational study evaluates the effect of therapy with cystic fibrosis transmembrane regulator (CFTR) modulators on CFTR function measured by the CFTR biomarker intestinal current measurement (ICM), nasal potential difference (NPD) and sweat chloride in a post-approval setting in patients with cystic fibrosis (CF).

DETAILED DESCRIPTION:
Cystic fibrosis transmembrane regulator (CFTR) biomarker (intestinal current measurement (ICM), nasal potential difference (NPD), sweat chloride) before the start of therapy and 12 and 52 weeks after initiation of therapy Clinical parameters (anthropometry, lung function, lung magnetic resonance imaging (MRI), lung computer tomography (CT)) before the start of therapy and after initiation of therapy Assessment of airway secretion specimens before the start of therapy and after initiation of therapy

ELIGIBILITY:
Inclusion Criteria:

* Decision for cystic fibrosis (CF) transmembrane regulator (CFTR)-modulator therapy by the patient and the caring CF physician
* Signed informed consent form (ICF) and, where appropriate, signed assent form.

Exclusion Criteria:

* Ongoing participation in an investigational drug study (including studies investigating lumacaftor, tezacaftor or ivacaftor)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cystic Fibrosis patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Intestinal current measurement (ICM) | 12 weeks
  Absolute change from baseline of the chloride secretory ion current induced by cyclic adenosine monophosphate (cAMP) stimulation (forskolin/3-isobutyl-1-methylxanthine (IBMX)) in rectal tissue determined by intestinal current measurement (ICM) as a cystic fibrosis transmembrane conductance regulator (CFTR) biomarker

SECONDARY OUTCOMES:
Forced expiratory volume in 1 second (FEV1) | 12, 52, 104 weeks
  Absolute change from baseline in percent predicted forced expiratory volume in 1 second (FEV1) in spirometry
Nasal potential Difference (NPD) | 12 weeks
  Absolute change from baseline total chloride response (zero chloride and isoproterenol) in nasal potential Difference (NPD) as a cystic fibrosis transmembrane conductance regulator (CFTR) biomarker
Sweat chloride | 12, 52, 104 weeks
  Absolute change from baseline of the chloride concentration in Gibson-Cooke pilocarpine iontophoresis sweat test as a cystic fibrosis transmembrane conductance regulator (CFTR) biomarker
Lung clearance index (LCI) | 12, 52, 104 weeks
  Absolute change from baseline of the lung clearance index (LCI)
Lung magnetic resonance imaging (MRI) | 12, 52, 104 weeks
  Absolute change from baseline in lung magnetic resonance imaging (MRI) score (Heidelberg MRI score ranging from 0 to 72 with higher values associated with worsening of the outcome; Eichinger et al. Eur J Radiol 2012)
Lung computer tomography | 52, 104 weeks
  Absolute change from baseline in lung computer tomography (CT) score (Brody score ranging from 0 to 40,5 with higher values associated with worsening of the outcome; Brody et al. J Thorac Imaging 2006)
Paranasal sinus magnetic resonance imaging (MRI) | 12, 52, 104 weeks
  Absolute change from baseline in paranasal sinus magnetic resonance imaging (MRI) score (Sinunasal MRI score ranging from 0 to 68 with higher values associated with worsening of the outcome; Sommerburg et al. Ann Am Thorac Soc 2020)
Fecal elastase | 12, 52, 104 weeks
  Absolute change from baseline in fecal elastase-1 (FE-1) levels
Weight | 12, 52, 104 weeks
  Absolute change from baseline in weight
Airway Microbiome | 4, 12, 52, 104 weeks
  Absolute change in shannon index representing the alpha-diversity in sputum samples
Sputum Elasticity | 4, 12, 52, 104 weeks
  Absolute change in the elastic modulus (G') in sputum samples measured with a rheometer
Sputum Viscocity | 4, 12, 52, 104 weeks
  Absolute change in the viscous modulus (G'') in sputum samples measured with a rheometer

CONTACTS AND LOCATIONS:
Overall Officials: Simon Y Graeber, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (4):
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Justus-Liebig-University Giessen, Giessen
  - Hannover Medical School, Hanover
  - University of Heidelberg, Heidelberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schaupp L, Addante A, Voller M, Fentker K, Kuppe A, Bardua M, Duerr J, Piehler L, Rohmel J, Thee S, Kirchner M, Ziehm M, Lauster D, Haag R, Gradzielski M, Stahl M, Mertins P, Boutin S, Graeber SY, Mall MA. Longitudinal effects of elexacaftor/tezacaftor/ivacaftor on sputum viscoelastic properties, airway infection and inflammation in patients with cystic fibrosis. Eur Respir J. 2023 Aug 3;62(2):2202153. doi: 10.1183/13993003.02153-2022. Print 2023 Aug. PMID 37414422
- [Derived] Graeber SY, Renz DM, Stahl M, Pallenberg ST, Sommerburg O, Naehrlich L, Berges J, Dohna M, Ringshausen FC, Doellinger F, Vitzthum C, Rohmel J, Allomba C, Hammerling S, Barth S, Ruckes-Nilges C, Wielputz MO, Hansen G, Vogel-Claussen J, Tummler B, Mall MA, Dittrich AM. Effects of Elexacaftor/Tezacaftor/Ivacaftor Therapy on Lung Clearance Index and Magnetic Resonance Imaging in Patients with Cystic Fibrosis and One or Two F508del Alleles. Am J Respir Crit Care Med. 2022 Aug 1;206(3):311-320. doi: 10.1164/rccm.202201-0219OC. PMID 35536314
- [Derived] Graeber SY, Vitzthum C, Pallenberg ST, Naehrlich L, Stahl M, Rohrbach A, Drescher M, Minso R, Ringshausen FC, Rueckes-Nilges C, Klajda J, Berges J, Yu Y, Scheuermann H, Hirtz S, Sommerburg O, Dittrich AM, Tummler B, Mall MA. Effects of Elexacaftor/Tezacaftor/Ivacaftor Therapy on CFTR Function in Patients with Cystic Fibrosis and One or Two F508del Alleles. Am J Respir Crit Care Med. 2022 Mar 1;205(5):540-549. doi: 10.1164/rccm.202110-2249OC. PMID 34936849